CLINICAL TRIAL: NCT06381960
Title: Clinical Study on the Prevention and Treatment of Postoperative Metastasis in Stage IIA-IIIA Lung Cancer With Negative Expression of Driver Genes by Fuzheng Quxie Recipe
Brief Title: Clinical Study on the Prevention and Treatment of Postoperative Metastasis of Lung Cancer by Fuzheng Quxie Recipe
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jianhui Tian (Other)
Responsible Party: Sponsor-Investigator, Jianhui Tian, professor, Shanghai Municipal Hospital of Traditional Chinese Medicine
Organization: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022LJ014
Record Dates: First submitted 2024-03-15; First posted 2024-04-24 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Chinese medicine placebo granules + regular chemotherapy; (Placebo Comparator): Control group
  Interventions: Drug: Fuzhengquye Fang Recipe simulant
- Daily Fuzheng Quxie Recipe granules + regular chemotherapy (Experimental): Treatment Group
  Interventions: Drug: Fuzheng Quxie Recipe

INTERVENTIONS:
Drug: Fuzheng Quxie Recipe — Treatment group: Fuzheng Quxie Recipe (Yifei Sanjie Recipe) ingredients: Sheng Huang Qi 15g, Jiao Bai Zhu 15g, Bai Fu Ling 15g, Bei Sha Shen 15g, Zhe Mai Dong 15g, Dang Shen 15g, Shu Yang Quan 15g, Xia Ku Cao 15g, Sheng Mu Li 15g, Shi Jian Chuan 15g, Shi Shang Bai 15g, and Hai Zao 15g. Combined with basic chemotherapy after lung cancer.
  Other Names: Fuzheng Quxie Formula；Yifei Sanjie Recipe；Yifei Sanjie Formula；
  Arms: Daily Fuzheng Quxie Recipe granules + regular chemotherapy
Drug: Fuzhengquye Fang Recipe simulant — Control group: Fuzhengquye Fang Recipe simulant, which was prepared into control group placebo drug according to 5% of the drug content in the treatment group. Combined with basic chemotherapy after lung cancer.
  Other Names: no other names
  Arms: Daily Chinese medicine placebo granules + regular chemotherapy;

SUMMARY:
To address the clinical challenge of postoperative metastasis in stage IIA-IIIA non-small cell lung cancer with negative driver gene expression, there is a lack of effective diagnostic and therapeutic measures. Based on this, investigators propose to carry out a clinical study on the prevention and treatment of postoperative metastasis of IIA-IIIA stage lung cancer with negative driver gene expression with the formula of supporting the positive and dispelling the evil.

DETAILED DESCRIPTION:
In this study, investigators actively explored the establishment of a combined Chinese and Western medicine prevention and treatment programme in response to the urgent clinical need for the lack of effective diagnostic and therapeutic options for postoperative patients with stage IIA-IIIA non-small cell lung cancer who are clinically negative for the expression of driver genes.

1. To objectively evaluate the efficacy of "Fuzheng Quxie Recipe" in preventing and treating postoperative metastasis in stage IIA-IIIA non-small cell lung cancer with negative expression of driver genes, including its effects on disease-free survival, quality of life, and regulation of immune function of the patients, by means of a clinical study in accordance with international standards;
2. To test the immunohistology, circulating tumour cells and tiny residual lesions of the patients, and to screen out the population with the advantages of Chinese medicine treatment. Based on this, investigators will establish an efficacy prediction model including the evaluation of peripheral immune function status and the expression level of circulating tumour cells, in order to improve the level of precision treatment after radical lung cancer surgery.
3. Through conducting high-level clinical research in line with international standards, obtaining high-level evidence-based medical evidence, screening the advantageous populations of Chinese medicine in treating lung cancer metastasis, and forming a standardised diagnostic and treatment plan/guidelines on Chinese medicine or international guidelines on combining traditional Chinese and Western medicines for the prevention and treatment of post-surgical metastasis of lung cancer that can be promoted and applied, so as to provide a solid scientific basis for the transformation of clinical results and the development of new medicines, and to promote the improvement of the efficiency of the prevention and control of lung cancer as a whole.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical stage IIA-IIIA lung adenocarcinoma after radical surgery (patients within 6 weeks after surgery);
2. Negative driver gene expression (no EGFR, ALK, ROS1 mutations) and PD-1/L1 expression <1%;
3. Meets the diagnostic criteria for Qi-Yin Deficiency Syndrome. The primary symptoms include cough, low sputum, shortness of breath, hoarseness, weakness, and thirst without wanting to drink. Secondary symptoms include spontaneous, night sweat, dysphoria in chestpalms-soles, red tongue or tooth-marked tongue, and a weak pulse. At least two primary symptoms and one of the secondary symptoms are present;
4. Patients aged between 18-75 years;
5. Patients with basically normal blood and biochemical indices, etc., without serious viral or bacterial infections; patients without organ failure and serious heart disease (blood bilirubin <68 μmol/L, aspartate aminotransferase <90 IU/L, creatinine <350 μmol/L, white blood cell count >3.5 × 109/L and less than 12 × 109/L, platelet count >80 × 109/L, and (erythrocyte pressure area >0.20);
6. Tumour PS score ≤2 and no other serious comorbidities;
7. The subjects themselves were well informed and agreed to participate in the study by signing an informed consent form and had good compliance;
8. Non-pregnant and lactating patients;
9. Passing the chemotherapy-related indexes;
10. No allergic reaction to the ingredients in the formula.

Exclusion Criteria:

1. Patients who are incompletely resected or whose cancer has undergone recurrence or metastasis;
2. Patients who are being treated with other drugs or therapies (including other Chinese herbal medicines, immunological drugs, radiotherapy, etc.);
3. Patients who are themselves mentally ill and have a lack of autonomous behaviour;
4. Women who are pregnant, preparing for pregnancy or breastfeeding;
5. Combined heart, lung, brain, liver, kidney and haematopoietic system and other serious diseases, psychiatric patients;
6. Allergic or known hypersensitivity to the components of the drug;
7. Patients who are participating in other clinical trials or have participated in other clinical trials within 3 months;
8. Alcohol and/or psychoactive substances abuse, drug abusers and dependent persons;
9. Other pathologies or conditions that, in the judgement of the investigator, have the effect of reducing the likelihood of enrolment or complicating enrolment, e.g., frequent changes in the work environment, unstable living conditions, and other conditions that predispose to loss of visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival, DFS | Checks were performed before the start of treatment and every 6 months after the procedure. Observational follow-up until 5 years postoperatively.
  Refers to the time between the start of randomisation and disease relapse or (for any reason) death. Imaging examination: chest CT examination before the beginning of treatment and every 6 months after the operation. Patients found to have recurrent metastases were discharged from the group for standardised treatment when the pathological diagnosis was clear. Observation and follow-up were carried out until 5 years after the operation, and the calculation of disease-free survival rate, disease-free survival period and median survival period were carried out.

SECONDARY OUTCOMES:
Overall survival,OS | The follow-up was observed until 5 years postoperatively, and overall and median survival calculations were performed.
  Endpoint indicator, defined as the time from the start of randomisation to death due to any cause.
Minimal residual disease, MRD | One test was performed before and 6 months after the intervention.
  Second-generation sequencing NGS method was used to detect MRD in peripheral blood of the study subjects to obtain a superior population screening model for TCM treatment.
Circulating Tumour Cell Assay | One test was performed before and 6 months after the intervention.
  Specimen collection method: 10ml of venous blood was taken from the patient's middle elbow vein with EDTA blood collection tube, and the blood collection tube was repeatedly reversed for mixing, and then centrifuged at 2000g for 10min, the supernatant was retained, and in order to further remove excess cellular components, it should be centrifuged again at 8000g for 10min.The separated plasma was frozen and stored at -80℃, or was extracted immediately according to the extraction kit instructions. The remaining blood cells were added to saline to replenish 10 ml and immediately isolated from circulating tumour cells.
Chinese Medicine Symptom Score | Recorded once before and once 6 months after the intervention, continuing for 18 months.
  According to the "Shanghai Municipal Chinese Medicine Disease Diagnosis and Treatment Routine", 10 Chinese medicine symptoms of cough, sputum, chest pain, chest tightness, shortness of breath, fatigue, loss of appetite, insomnia, dry mouth and throat and spontaneous sweating were observed, with severity scored according to 0-3, and were recorded once before the intervention and once 6 months after the intervention. Significant effect: the reduction of TCM symptom scores was greater than or equal to 70% after the intervention; Effective: the reduction of TCM symptom scores was greater than or equal to 30% and less than 70% after the intervention; Ineffective: the reduction of TCM symptom scores was less than 30% after the intervention or higher than before.
Quality of life assessment | Recorded once before and once 6 months after the intervention, continuing for 18 months.
  The Quality of Survival Scale for Lung Cancer Patients EORTC QLQ-LC43 was used, which consists of EORTC QLQ-C30 (core scale) and EORTC QLQ-LC13 Th (characteristic subscale of lung cancer). It mainly scores lung cancer patients on 5 domains related to functioning, general clinical symptoms, characteristic sub-symptoms, general health status and financial difficulties, and is recorded once before and 6 months after the intervention. The score ranges for each of these five areas lie on a scale of 0-100. Higher scores on the function-related domains indicate poorer functioning of the organism; higher scores on the general clinical symptoms and characteristic sub-symptoms indicate more severe symptoms; higher scores on the general health status indicate better status; and higher scores on the economic hardship status indicate more financial hardship.
Cellular immunity (CD3） | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
Cellular immunity (CD4) | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
Cellular immunity (CD8) | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
Cellular immunity (CD16) | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
Cellular immunity (CD56） | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
regulatory T cells | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
myeloid-derived suppressor cells （MDSCs） | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
natural killer （NK）cells | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
IL-1 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
IL-2 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
IL-6 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
IL-8 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
IL-10 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Immunological indicators
CEA | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Tumour marker
CA125 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Tumour marker
CA153 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Tumour marker
Cyfra21-1 | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Tumour marker
SCC | The test was performed once before the intervention and once 6 months after the intervention,continuing for 18 months.
  Tumour marker
Peripheral blood systemic immunoinflammatory index | The test was performed once before the intervention and once 6 months after the intervention, continuing for 18 months.
  SII=peripheral blood platelet count (x10/L) x peripheral blood neutrophil count (x10/L)/peripheral blood lymphocyte count (x10%/L).
  PNI:serum albumin(g/L)+lymphocyte count(10/L)x5. The critical value was calculated according to the ROC curve, and according to the critical value, the above indexes were classified into high level group and low level group.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhui Tian, professor, Study Director — Shanghai University of Traditional Chinese Medicine
Locations (5):
- China (5):
  - Shanghai Chest Hospital, Changning, Shanghai Municipality
  - Shanghai General Hospital, Hongkou, Shanghai Municipality
  - Shanghai Traditional Chinese Medicine-Integrated Hospital, Hongkou, Shanghai Municipality
  - Shanghai Municipal Hospital of Traditional Chinese Medicine, Jing’an, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Yangpu, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu F, Yang Y, Luo Y, Luo B, Yao J, Zhou Y, Li M, Wu J, Shi W, Jiang L, Huang Q, Fang W, Fang Z, Li Y, Tian J. Efficacy of Fuzheng Quxie Formula Against Postoperative Metastasis of Lung Cancer in Stage IIA-IIIA With Negative Driver Genes: Protocol for a Multicenter, Double-Blind, Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 24;14:e66342. doi: 10.2196/66342. PMID 41135941

DOCUMENTS (2):
  • Study Protocol (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT06381960/Prot_000.pdf
  • Informed Consent Form (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT06381960/ICF_001.pdf